CLINICAL TRIAL: NCT02884037
Title: Could Rifaximin Modify the Pathogenesis of NAFLD? AMulticenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Rifaximin Modify the Pathogenesis of Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nasser Mousa, Prof of Tropical Medicine and Hepatology, Mansoura University
Other Study IDs: R/16.02.80
Record Dates: First submitted 2016-07-29; First posted 2016-08-30 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; Rifaximin; Endotoxin and Homeostatic Model Assessment
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Rifaxmin group
  Interventions: Drug: Rifaximin group 1
- 2: placebo group

INTERVENTIONS:
Drug: Rifaximin group 1 — Rifaximin: 1100mg/day, 550 mg tablets 1 × 2 before meals
  Groups: 1

SUMMARY:
In this multicentric, double-blind, randomized,placebo-controlled study, the investigators hypothesized that rifaximin might act on Gram-negative bacteria and intestinal bacterial overgrowth(IBO) thereby inhibiting lipopolysaccharides(LPS)-mediated proinflammatory cytokine production. This work evaluates the efficacy of 6 months administration of rifaximin in NAFLD patients.

DETAILED DESCRIPTION:
The investigators aimed to study the effect of rifaximin on NASH. 50 patients with biopsy-proven NASH were enrolled in this double-blind, randomized,placebo-controlled study. BMI, AST, ALT, gamma glutamyl transferase (γ-GGT), lipid profile, homeostatic model assessment (HOMA), serum endotoxin, Toll-like receptor 4 (TlR4), interleukin-6 (IL-6), IL-10, tumor necrosis factor-α (TNF-α) and cytokeratin-18 (CK-18) levels were measured before and after a 6 month administration of rifaximin (1100mg/day, 550 mg tablets 1 × 2 before meals).

ELIGIBILITY:
Inclusion Criteria:

1. women or men aged 18-65 years.
2. biopsy-proven NASH without or with mild to moderate fibrosis (fibrosis stage 0-3)in the preceding year.
3. persistently abnormal ALT on 2 occasions.
4. participants have provided written informed consent before screening.
5. all patients counseled about the standard of care treatment (e.g., diet andexercise).
6. Strict requirements for weight stability between the time of biopsy and study entry.

Exclusion Criteria:

1. Cirrhotic NAFLD (METAVIR stage 4).
2. Combined viral hepatitis B and C infection.
3. increased alcohol intake (>20 g/day) and hypothyroidism.
4. co-existence of another type of biliary tract or pancreatic or liver diseases
5. lactating or pregnant women.
6. allergy to rifamycin or rifaximin.
7. systemic inflammatory conditions (e.g. Connective tissue diseases and inflammatory bowel diseases).
8. bariatric surgery and blind loop.
9. evidence of hepatic decompensation (ascites, hepatic encephalopathy, and varices),
10. history of myocardial infarction and/ or stroke within 6 months.
11. drugs that alter the gut flora e.g. Lactulose, systemic antibiotic, cholestyramine within three months, (l) cancers especially HCC, and (m)patients with renal impairment (estimated GFR <60ml/min/1.73m2).

(n) Major dose change orintiation of biguanides, metformin, thiazolidinediones, insulin, fibrates, statins, and anti-obesity medications within three months before the onset of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this multicentric, double-blind, randomized,placebo-controlled study, we enrolled consecutively 1072 participants with hepatitis irrespective to their etiologies referred to the Tropical Medicine and Internal Medicine Departments (Mansoura University), Tropical Medicine Department (Zagazig University), and Internal Medicine and Endemic Diseases and Gastroenterology Departments (Aswan University)from May 2012 to October 2016. All participants underwent to the following appraisal: physical and biochemical examination, complete history taking, abdominal ultrasound, and percutaneous ultrasound liver biopsy.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
serum ALT | 6 months
  U/l
serum endotoxins | 6 months
  EU/ml
TLR-4 | 6 months
  ng/ml

SECONDARY OUTCOMES:
Fasting Glucose | 6 months
  mg/dl
, Insulin, | 6 months
  μIU/ml
CK-18,TNF-α, IL-6, IL 10 | 6 months
  pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser H Mousa,MD,mousa_medic@yahoo.com. +201227029213, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No